CLINICAL TRIAL: NCT06038422
Title: Clinical Study on Efficacy and Safety of GTP Regimen in the Treatment of Refractory/Recurrent Hemophagocytic Lymphohistiocytosis
Brief Title: GTP Regimen in the Treatment of Refractory/Recurrent HLH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, director of department, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20230717001
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Refractory; Recurrence; Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Recurrence; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GTP regimen treated patients (Experimental): R/R HLH patients treated with GTP regimen
  Interventions: Drug: GTP regimen

INTERVENTIONS:
Drug: GTP regimen — Refractory/recurrent hemophagocytic lymphohistiocytosis patients will be treated with GTP regimen (Emapalumab+Teniposide+Methylprednisolone)

SUMMARY:
The goal of this clinical trial is to learn about efficacy and safety of GTP regimen in refractory/recurrent hemophagocytic lymphohistiocytosis. The main questions it aims to answer are:

* Overall remission rate of GTP regimen in R/R HLH
* Adverse effect of GTP regimen Participants will be treated with GTP regimen

DETAILED DESCRIPTION:
Refractory/recurrent hemophagocytic lymphohistiocytosis will be treated with emapalumab combined with teniposide and methylprednisolone. Observed the overall response rate and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥1 month of age with HLH
2. Definitive diagnosis of HLH: meets the molecular diagnosis of pHLH or has a family history of HLH, or meets at least 5 of the 8 diagnostic criteria of HLH-2004.
3. The investigators assessed the presence of refractory/recurrent HLH disease. Patients must meet one of the following criteria assessed by the investigator:

   * Previous conventional HLH treatment did not respond.
   * The patients were not satisfied with the efficacy of conventional HLH treatment or their condition worsened.
   * HLH reactivation occurs. Reactivation is defined as: worsening of two or more HLH clinical and laboratory criteria (after initial remission).
4. According to the researchers, the expected survival was more than 2 weeks.
5. The informed consent is signed by the patient or his legal guardian (patients under 18 years), or by the patient's legally authorized representative.
6. Women who are fertile are willing to use a highly effective contraceptive method from the start of the study until 6 months after the end of the last course of treatment.

Exclusion Criteria:

1. There is active mycobacterium, histoplasma capsulatus, Salmonella, or leishmania infection.
2. There is uncontrolled active gastrointestinal bleeding.
3. The investigator believes that there are any serious comorbidities or any other conditions that make the patient unsuitable for treatment.
4. A history of hypersensitivity or hypersensitivity to any component of the drug in the study protocol, such as polysorbate.
5. Had received the BCG vaccine within 12 weeks prior to screening.
6. Have received live or attenuated vaccine (except BCG) within 4 weeks prior to screening.
7. Pregnancy patients.
8. Within 4 weeks prior to enrollment in this study, another concurrent clinical intervention study was enrolled.
9. There is any condition or circumstance that the investigator believes may cause the patient to be unable to complete the study or to comply with study procedures or requirements.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Overall remission rate